CLINICAL TRIAL: NCT04984577
Title: Phase II Trial of Compound Edaravone Injection for Treatment of Acute Ischemic Stroke -- a Multi-center, Randomized, Double-blind, Parallel, Multi-doses and Active-controlled Study
Brief Title: Study of Compound Edaravone Injection for Treatment of Acute Ischemic Stroke
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic realignment of sponsors.
Sponsor: Nanjing Yoko Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NJYK-CPEDRV-II
Record Dates: First submitted 2021-07-29; First posted 2021-07-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Compound Edaravone Injection-Low dose (Experimental)
  Interventions: Drug: Compound Edaravone Injection-Low dose
- Compound Edaravone Injection-High dose (Experimental)
  Interventions: Drug: Compound Edaravone Injection-High dose
- Edaravone Injection (Active Comparator)
  Interventions: Drug: Edaravone Injection
- Placebo Injection (Placebo Comparator)
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Compound Edaravone Injection-Low dose — Compound Edaravone Injection 30mg/dose (Edaravone 30mg, Taurine 600 mg), one dose every 12 hours, continue for 14 days
  Arms: Compound Edaravone Injection-Low dose
Drug: Compound Edaravone Injection-High dose — Compound Edaravone Injection 50mg/dose (Edaravone 50mg, Taurine 1000 mg), one dose every 12 hours, continue for 14 days
  Arms: Compound Edaravone Injection-High dose
Drug: Edaravone Injection — Edaravone Injection 30mg/dose, one dose every 12 hours, continue for 14 days
  Arms: Edaravone Injection
Drug: Placebo injection — Placebo injection, one dose every 12 hours, continue for 14 days
  Arms: Placebo Injection

SUMMARY:
The primary objective of the study is to confirm the efficacy of compound Edaravone Injection via intravenous infusion every 12 hours in the patients with Acute Ischemic Stroke(AIS) in a double-blind, active-controlled manner. The study is also to examine the safety of compound Edaravone Injection for the AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients, diagnosed of ischemic stroke;
* Onset of stroke is less than or equal to 48 hours;
* There are clear signs of neurological deficit: 4≤NIHSS score≤24, and also, the sum of NIHSS score for the upper limb and the lower limb is greater than or equal to 2;
* Patients signed written inform consent

Exclusion Criteria:

* Cranial CT scan finds intracranial bleeding disorders: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage;
* Iatrogenic stroke;
* Severe disturbance of consciousness: NIHSS category 1a for consciousness is greater than 1；
* The mRS score prior to this onset is greater than 1;
* Transient ischemic attack (TIA);
* SBP after blood pressure control is still greater than or equal to 220 mmHg, or DBP after blood pressure control is still greater than or equal to 120 mmHg;
* Patients with severe mental disorders and dementia;
* ALT or AST is greater than 2.0×ULN; Serum Creatinine (SCr) is greater than 1.5×ULN or Creatinine Clearance (CrCl) is less than 50 ml/min;
* Therapeutic neuroprotective agents have been applied after onset of stroke, including commercially available edaravone, nimodipine, ganglioside, citicoline, piracetam, butyl benzene peptides, Urinary Kallidinogenase;
* Thrombectomy or interventional therapy has been applied or planned after this onset;
* Patients with malignant tumors or receiving concurrent antitumor treatment;
* Patients with severe systemic disease, life expectancy is less than 90 days;
* Allergic to edaravone , taurine or related excipients;
* Pregnant or lactating women;
* Have major surgery within 4 weeks before enrollment and not recovered enough to start the study;
* Participated in other clinical studies within 30 days before randomization;
* The investigators consider the patients are not suitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with mRS ≤1 on day 90 | day 90

SECONDARY OUTCOMES:
Changes of NIHSS score from baseline on day 14 | day 14
The proportion of patients with mRS ≤2 on day 90 | day 90
The proportion of patients with NIHSS score 0-1 (including motor function) on day 14, 30, 90 | day 14, 30, 90
The proportion of patients with ADL-BI ≥95 on day 14, 30, 90 | day 14, 30, 90
EQ-5D score on day 90 | day 90
Ordinal Distribution of mRS on day 90 | day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital，Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No